CLINICAL TRIAL: NCT07057817
Title: Randomised Controlled Trial Comparing Partial Calcanectomy Plus Local Application Antibiotic Impregnated Bone Graft Substitute for Calcaneal Osteomyelitis vs Partial Calcanectomy Alone (The ACHILLS Trial)
Brief Title: The ACHILLS Trial; Application of Cerament in Heel Infection for Lower Limb Salvage
Acronym: ACHILLS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCSI-ACHILLS
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Osteomyelitis; Diabetes; Calcanectomy
Keywords: Calcanectomy; Eq5d5l
MeSH Terms: conditions — Osteomyelitis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Calcanectomy with Cerament G (Experimental): Patients will undergo partial calcanectomy with the application of Cerament G.
  Interventions: Device: Cerament G
- Standard Partial Calcanectomy (Active Comparator): Patients will undergo partial calcanectomy with standard antibiotic therapy.
  Interventions: Other: Standard Surgical Managment

INTERVENTIONS:
Device: Cerament G — Partial Calcanectomy plus cerament G
  Arms: Partial Calcanectomy with Cerament G
Other: Standard Surgical Managment — Partial Calcanectomy as standard of care
  Arms: Standard Partial Calcanectomy

SUMMARY:
The ACHILLS Trial is a multicentre randomised controlled feasibility study comparing partial calcanectomy with and without the use of an antibiotic-impregnated bone graft substitute (Cerament G) for treating calcaneal osteomyelitis, specifically on wound healing rates, re-infection, and overall efficacy in a sample of 30 patients over a one-year period.

DETAILED DESCRIPTION:
Calcaneal osteomyelitis is a severe infection of the heel bone, frequently linked to peripheral arterial disease and diabetes, which complicates the healing process. This condition can lead to chronic wounds, persistent pain, and, in extreme cases, the need for limb amputation. Standard treatment often involves partial or total calcanectomy, where the infected bone is surgically removed, significantly impacting patients' mobility and quality of life.

The ACHILLS Trial is a multicentre, randomised controlled feasibility study designed to assess the efficacy of partial calcanectomy with and without the use of Cerament G, an antibiotic-impregnated bone graft substitute.

The primary objective is to determine the rate of wound healing in patients undergoing partial calcanectomy for osteomyelitis who receive Cerament G.

Secondary objectives include assessing time to wound healing, rates of re-infection, hospital stay duration, need for extended antibiotic therapy, financial impact, and overall quality of life.

The trial will involve 30 participants, aged 18 and older, undergoing partial calcanectomy for osteomyelitis. Participants will be randomly assigned to one of two groups: one receiving partial calcanectomy with Cerament G, and the other receiving partial calcanectomy alone with standard antibiotic therapy. The study will monitor patients for one year, with data collected at multiple intervals to monitor wound healing, re-infection rates, and other outcomes.

Cerament G, comprising calcium sulphate and hydroxyapatite, serves as a bone substitute and delivers a localised antibiotic (gentamycin) directly to the infection site. This approach aims to reduce infection rates, promote bone healing, and minimise the need for further surgical interventions.

The results from this feasibility study may result in a larger trial, potentially leading to improved management strategies for calcaneal osteomyelitis, reduced healthcare costs, and enhanced patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Undergoing partial calcanectomy
* Patients with Type1 or Type 2 Diabetes
* Patients will be stratified by Pulse status and eGFR

Exclusion Criteria:

* Patients unfit for surgery
* Patients unable to provide informed consent
* Patients with overwhelming sepsis that require major amputation
* Patients with hypersensitivity to aminoglycosides
* Pre-existing calcium metabolism disorder
* Severe renal impairment
* Patients in whom major limb amputation is deemed inevitable by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound Healing | 1 months post-surgery
  To determine the number of patients achieving complete wound healing in patients undergoing treatment with cerament G compared to those with partial calcanectomy alone by measuring wound volume
Rate of Wound Healing | 3 months post-surgery
  To determine the number of patients achieving complete wound healing in patients undergoing treatment with cerament G compared to those with partial calcanectomy alone by measuring wound volume
Rate of Wound Healing | 6 months post-surgery
  To determine the number of patients achieving complete wound healing in patients undergoing treatment with cerament G compared to those with partial calcanectomy alone by measuring wound volume
Rate of Wound Healing | 12 months post-surgery
  To determine the number of patients achieving complete wound healing in patients undergoing treatment with cerament G compared to those with partial calcanectomy alone by measuring wound volume

SECONDARY OUTCOMES:
Time to Wound Healing | 1, 3, 6, and 12 months post-surgery
  Number of days taken to achieve full wound healing.
Quality of life measured with the EQ5D5L (Health Questionnaire) | 1 month post-surgery
  Impact on patients quality of life measured using the EQ-5D-5L health questionnaire. The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Quality of life measured with the EQ5D5L (Health Questionnaire) | 3 months post-surgery
  Impact on patients quality of life measured using the EQ-5D-5L health questionnaire, The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Quality of life measured with the EQ5D5L (Health Questionnaire) | 6 months post-surgery
  Impact on patients quality of life measured using the EQ-5D-5L health questionnaire, The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Quality of life measured with the EQ5D5L (Health Questionnaire) | 12 months post-surgery
  Impact on patients quality of life measured using the EQ-5D-5L health questionnaire
Cost to Patients Questionaire (CoPaQ) | 12 months post-surgery
  Measures patients' and caregivers' out-of-pocket expenses (e.g., travel) and indirect costs (e.g., loss of income). It is divided into two sections 1. Costs for Patients Questionnaire and 2. Sociodemographic and Health Questions..
Length of Hospital Stay | 12 months post-surgery
  Length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: James Walsh, Principal Investigator — Beaumont Hospital
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No